CLINICAL TRIAL: NCT01213862
Title: Home Visit Impact on Knowledge of Disease, Self-Care Skills and Quality of Life of Heart Failure Patients: Randomized Clinical Trial
Brief Title: Home Based Intervention Led by Nurse in Brazil
Acronym: HFHELENI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Principal Investigator, Eneida Rejane Rabelo da Silva, Professor, PhD., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGS and HCPA 09111
Record Dates: First submitted 2009-11-09; First posted 2010-10-04 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Heart Failure
Keywords: Home Based education; Knowledge of Disease; Self-Care Skills; Quality of Life; Heart Failure; Randomized Clinical Trial
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention and control (Experimental): * Group I - Intervention: Routine follow-up in a reference health institution with four home visits and four telephone contacts with specialist nurses.
  * Group II - Control: Routine follow-up with the health team in the reference institution.
  Interventions: Behavioral: Home Based Education

INTERVENTIONS:
Behavioral: Home Based Education — There will provided education about what is heart failure, its causes, how to recognize signs and symptoms, monitoring of weight and blood pressure, the importance of compliance to treatment. Patients will be instructed about the medications; a guide to rest and exercise, sexual activity, vaccines, travel and diet will be provided. The involvement of the family will be encouraged; the contact with the team should be done when: patient observes an increase of 1 or 2 kg of weight in 2-3 days, worsening of dyspnea on effort, edema in legs / abdomen, worsening of cough, persistent vomiting, syncope, sputum with blood, fever, persistent tachycardia. In phone calls made between home visits, the compliance to treatment will be evaluated and reinforced.
  Other Names: Education on Heart Failure; Home based intervention

SUMMARY:
Home visits (HV) are one of the multidisciplinary approaches that has already shown to benefit the follow-up of Heart Failure (HF) patients. It is considered to be one of the most effective and humane approaches as it educates and takes care of the patient in his/her routine environment. In this study, the follow-up of HF patients in a home setting after being discharged from hospital will include the reinforcement, monitoring and re-evaluation of guidelines previously provided about the disease and self-care, compliance to prescribed medicines and, specially, the early recognition of decompensation signs and symptoms by patients and their caregivers.

DETAILED DESCRIPTION:
The epidemiological overview of cardiovascular diseases in which HF turns out to be the main cause of re-hospitalizations in the Unified Health System, which has not changed over the years, impairs the management of the limited resources of the public health system. Additionally, HF leads to substantial damage to the quality of life of patients, many of them at a socially productive age, resulting in early retirements and absences. In this study, the objective is to evaluate the impact of the follow-up of heart failure patients at home, interspersed with telephone contacts, by the nursing team, after hospital discharge, regarding knowledge of the disease, self-care skills and quality of life improvement, compared with the conventional follow-up of patients in a 6-month period without this intervention, as well as to build a mobile-technology computer structure to make the use of cardiology nursing evaluation forms viable; correlate sociodemographic and clinical characteristics with treatment compliance and re-hospitalization rates in both; and ascertain home follow-up costs.

With this purpose, a two-center randomized clinical trial, blinded for the endpoints re-hospitalization and costs, was designed.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Age equal to or above 18 years
* Diagnosis of heart failure with systolic dysfunction (ejection fraction ≤ 45%)
* Hospitalized for heart failure decompensation and who agree to participate in the study by signing a Free Informed Consent Form.

Exclusion Criteria:

* Patients presenting with communication barriers and suffering from degenerative neurological diseases.
* Patients who had Acute Coronary Syndrome (ACS) in the past 6 months before randomization
* Patients with renal/hepatic/pulmonary or systemic disease who may confuse the interpretation of findings or result in limited life expectancy
* Surgical or therapeutic treatment that may influence the follow-up
* Pregnancy
* Diagnosis of Heart Failure secondary to:

  * sepsis
  * myocarditis
  * acute myocardial infarction
  * peripartum cardiomyopathy and other acute cause
* No interest in receiving home visits
* Living more than 10 km away for the original hospital
* No possibility of telephone contact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Knowledge of the disease | Home visit 7 days after discharge
  This primary outcome will be measured at each home visit, which will have different intervals, according to the research protocol.
Self-care skills. | Home visit 7 days after discharge.
  This primary outcome will be measured at each home visit, which will have different intervals, according to the research protocol.
Quality of Life | Home visit 7 days after discharge
  This primary outcome will be measured at each home visit, which will have different intervals, according to the research protocol.

SECONDARY OUTCOMES:
Changes in functional class. | Home visits (HV) starting 7days after discharge.
  This secundary outcome will be measured at each visit and phone call, which will have different intervals, according to the research protocol.
Presentation to emergency department | Home visits starting 7 days after discharge.
  This secundary outcome will be measured at each visit and phone call, which will have different intervals, according to the research protocol.
Compliance score. | Home visits starting 7 days after discharge.
  This secundary outcome will be measured at each visit and phone call, which will have different intervals, according to the research protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo da Silva, RN, ScD, Principal Investigator — Federal University of Rio Grande do Sul; Eneida R Rabelo da Silva, RN, ScD, Principal Investigator — Universidade Federal do Rio do Sul

REFERENCES:
- [Derived] Mussi CM, Ruschel K, de Souza EN, Lopes AN, Trojahn MM, Paraboni CC, Rabelo ER. Home visit improves knowledge, self-care and adhesion in heart failure: Randomized Clinical Trial HELEN-I. Rev Lat Am Enfermagem. 2013 Jan-Feb;21 Spec No:20-8. doi: 10.1590/s0104-11692013000700004. English, Portuguese. PMID 23459887